CLINICAL TRIAL: NCT02438605
Title: Dynamic CT Imaging After Nellix Endoprosthesis Implantation
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, M.D., PhD., Rijnstate Hospital
Other Study IDs: StM 596
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Aortic Aneurysm
Keywords: Nellix; EVAS; EVAR; Dynamic CT; Dyna CT
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment group: Patients eligible for AAA repair using Nellix and willing to participate in this trial.
  Interventions: Device: Nellix

INTERVENTIONS:
Device: Nellix

SUMMARY:
The Nellix Endovascular Sealing Prosthesis (EVAS) endoprosthesis is a new device aimed at prophylactic treatment of abdominal aortic aneurysms. In regular follow up conventional CT-imaging is used for surveillance. In this study dynamic CT imaging in patients pre- and post-operative will be assessed for device changes and anatomical variances.

ELIGIBILITY:
Inclusion Criteria:

* Nellix implantation

Exclusion Criteria:

* Use of chimneys or combined with other stent graft material

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients eligible for endovascular aortic repair using the Nellix endovascular sealing system
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in aortic aneurysm morphology as seen on dynamic CT after EVAS | 1 month

SECONDARY OUTCOMES:
Dynamic changes in neck morphology after EVAS | 1 month
Dynamic changes in common iliac artery morphology after EVAS. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands